CLINICAL TRIAL: NCT03081715
Title: Safety and Activity of Programmed Cell Death-1 Knockout Engineered T Cells in Patients With Previously Treated Advanced Esophageal Squamous Cell Carcinoma: An Open-label, Single-arm Phase 1 Study
Brief Title: PD-1 Knockout Engineered T Cells for Advanced Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Cancer Hospital (Other)
Collaborators: Anhui Kedgene Biotechnology Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Shixiu Wu, Professor, Hangzhou Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangzhouCH07
Record Dates: First submitted 2017-03-11; First posted 2017-03-16 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; immune checkpoint; PD-1; CRISPER; autologous cell infusion
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Masking Description: open-label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death 1(PD-1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and reinfused back into patients. To avoid allergic reactions, 50 mg hydrocortisone was intravenously injected into the patient 30 min before cells infusion every time. Best supportive care was also provided for patients.
  A total of 1 to 10 x 10^9 PD-1 Knockout T cells will be infused each cycle. Patients continued receiving treatment unless they had unacceptable adverse effects, or progressive disease confirmed by CT or they withdrew consent.
  Interventions: Other: PD-1 Knockout T Cells

INTERVENTIONS:
Other: PD-1 Knockout T Cells — Programmed cell death 1(PD-1) gene will be knocked out by CRISPR Cas9

SUMMARY:
This study will evaluate the safety of PD-1 knockout engineered T cells in treating advanced esophageal cancer. Blood or tissue samples will also be collected for research purposes.

DETAILED DESCRIPTION:
This is a prospective clinical study of ex-vivo selected, engineered, and expanded PD-1 knockout T cells from autologous origin. 16 advanced esophageal cancer patients are planned to receive two cycles of PD-1 knockout engineered T cells infusion. Immunological markers are analyzed as well.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or metastatic esophageal cancer
* Measurable disease
* Progressed after standard treatments
* ECOG performance status of 0-2
* Expected life span: >= 3 months
* Toxicities from prior treatment has resolved or ≤ grade 1
* Major organs function normally
* Women at pregnant ages should be under contraception
* Willing and able to provide informed consent

Exclusion Criteria:

* Other malignancy within 5 years prior to entry into the study, expect for treated non-melanoma skin cancer and cervical carcinoma in situ
* Poor vasculature
* Disease to the central nervous system
* Blood-borne infectious disease, e.g. hepatitis B
* History of mandatory custody because of psychosis or other psychological disease inappropriate for treatment deemed by treating physician
* With other immune diseases, or chronic use of immunosuppressants or steroids
* Pregnancy (women of childbearing potential:Refusal or inability to use effective means of contraception)
* Breastfeeding
* Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Response Rate | 1-3 months
  Response will be evaluated according to RECIST v1.1

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 months
  Number of participants with Adverse Events and grade as a measure of safety and tolerability of PD-1 knockout T cells using CTCAE v4.03

OTHER OUTCOMES:
Progression free survival (PFS) | 1 year
  From date of randomization until the date of first documented progression or date of death from any cause
Overall Survival (OS) | 1 year
  The time from randomization to death from any cause
Peripheral blood T lymphocyte subsets | 6 weeks
  Sera were collected at baseline and after the first cycle to measure T lymphocyte subsets with flow cytometry
Tumor-infiltrating T cells | Baseline and after treatment
  Baseline and post-treatment tissue samples were tested for the tumor-infiltrating T cells with immunofluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: shixiu wu, Professor, Principal Investigator — Hangzhou Cancer Hospital
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Niu Y, Shen B, Cui Y, Chen Y, Wang J, Wang L, Kang Y, Zhao X, Si W, Li W, Xiang AP, Zhou J, Guo X, Bi Y, Si C, Hu B, Dong G, Wang H, Zhou Z, Li T, Tan T, Pu X, Wang F, Ji S, Zhou Q, Huang X, Ji W, Sha J. Generation of gene-modified cynomolgus monkey via Cas9/RNA-mediated gene targeting in one-cell embryos. Cell. 2014 Feb 13;156(4):836-43. doi: 10.1016/j.cell.2014.01.027. Epub 2014 Jan 30. PMID 24486104
- [Background] Rosenberg SA, Restifo NP. Adoptive cell transfer as personalized immunotherapy for human cancer. Science. 2015 Apr 3;348(6230):62-8. doi: 10.1126/science.aaa4967. PMID 25838374
- [Background] Sharma P, Allison JP. Immune checkpoint targeting in cancer therapy: toward combination strategies with curative potential. Cell. 2015 Apr 9;161(2):205-14. doi: 10.1016/j.cell.2015.03.030. PMID 25860605